CLINICAL TRIAL: NCT00787579
Title: Assessment of Bifocal and Prismatic Bifocal Spectacles for Myopia Control in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Collaborators: Queensland University of Technology (Other)
Responsible Party: Desmond Cheng, Essilor International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Essilor
Record Dates: First submitted 2008-11-04; First posted 2008-11-07 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Myopia
Keywords: Myopia, bifocal, children
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bifocal spectacles (Active Comparator)
  Interventions: Device: Bifocal spectacles
- Prismatic bifocals (Active Comparator)
  Interventions: Device: Prismatic bifocal spectacles
- Single vision spectacles (No Intervention)

INTERVENTIONS:
Device: Bifocal spectacles — +1.50D bifocal spectacles
  Arms: Bifocal spectacles
Device: Prismatic bifocal spectacles — +1.50D bifocal spectacles combined with 3Δ base-in prisms
  Arms: Prismatic bifocals

SUMMARY:
1. To determine if the effect of near-addition lenses (bifocals) is more prominent for children with high myopia progression.
2. To study how different subject characteristics such as age, gender, baseline degree of myopia, baseline near phoria and baseline lag of accommodation affect the efficacy of bifocal lens wear in myopic children.
3. To investigate the effect of incorporating near base-in prisms along with the near-addition lenses (prismatic bifocals) on myopia progression in myopic children.

ELIGIBILITY:
Inclusion Criteria:

* Age: 8 to 13 years
* Myopia: -1.00 to -5.00 D
* Myopia progression: at least 0.50 D/yr
* Astigmatism and anisometropia: not more than 1.50 D
* Distance monocular visual acuity: 6/6 or better
* Near monocular visual acuity: 0.4 M or better
* Stereoacuity: not more than 40 sec of arc at 40 cm

Exclusion Criteria:

* Strabismus
* Ocular diseases

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2003-04; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Myopia progression, measured by cycloplegic autorefraction | Every 6 months

SECONDARY OUTCOMES:
Axial length, measured by A-scan ultrasonography | Every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Cheng, OD, MSc, Principal Investigator — Queensland University of Technology
Locations (1):
- Dr. Desmond Cheng & Associates, Mississauga, Ontario, Canada

REFERENCES:
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645
- [Derived] Cheng D, Woo GC, Drobe B, Schmid KL. Effect of bifocal and prismatic bifocal spectacles on myopia progression in children: three-year results of a randomized clinical trial. JAMA Ophthalmol. 2014 Mar;132(3):258-64. doi: 10.1001/jamaophthalmol.2013.7623. PMID 24435660
- [Derived] Cheng D, Schmid KL, Woo GC, Drobe B. Randomized trial of effect of bifocal and prismatic bifocal spectacles on myopic progression: two-year results. Arch Ophthalmol. 2010 Jan;128(1):12-9. doi: 10.1001/archophthalmol.2009.332. PMID 20065211